CLINICAL TRIAL: NCT05401916
Title: Efficacy of Intravenous Ibuprofen and Paracetamol on Postoperative Pain and Tramadol Consumption in Shoulder Surgery: Prospective, Randomized, Double-Blind Clinical Trial
Brief Title: Efficacy of Intravenous Ibuprofen and Paracetamol on Postoperative Pain and Tramadol Consumption in Shoulder Surgery
Acronym: Ibuprofen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Muhittin Calim, Principal Investigator, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: muhittincalim2
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain Management
Keywords: Postoperative pain; Intravenous ibuprofen; Intravenous paracetamol; Shoulder surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol; Analgesia, Patient-Controlled; Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized Double Blind Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous paracetamol (Active Comparator): Intravenous paracetamol 1 g paracetamol will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received Tramadol with intravenous patient controlled analgesia (IV PCA) pump during postoperative 24 hours. The PCA solution will be prepared with 500 mg tramadol in 100 mL of saline (5 mg/ml). The PCA device was adjusted as infusion: 2 ml/h, bolus: 2 ml, lockout period: 15 min.
  Interventions: Drug: Tramadol; Drug: Paracetamol
- Intravenous ibuprofen (Active Comparator): 800 mg ibuprofen (diluted with 250 ml saline) will be administered 30 minutes before the end of surgery.
  All administrations will be applied through IV infusion over 30 minutes. Patients will be received Tramadol with intravenous patient controlled analgesia (IV PCA) pump during postoperative 24 hours. The PCA solution will be prepared with 500 mg tramadol in 100 mL of saline (5 mg/ml). The PCA device was adjusted as infusion: 2 ml/h, bolus: 2 ml, lockout period: 15 min.
  Interventions: Drug: Tramadol; Drug: Ibuprofen

INTERVENTIONS:
Drug: Tramadol — Patients will be received tramadol with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 500 mg tramadol in 100 mL of saline (5 mg/ml). The PCA device was adjusted as infusion: 2 ml/h, bolus: 2 ml, lockout period: 15 min.
  Other Names: Intravenous patient-controlled analgesia
Drug: Paracetamol — 1 g paracetamol will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received tramadol with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 500 mg tramadol in 100 mL of saline (5 mg/ml). The PCA device was adjusted as infusion: 2 ml/h, bolus: 2 ml, lockout period: 15 min.
  Other Names: Intravenous paracetamol
  Arms: Intravenous paracetamol
Drug: Ibuprofen — 800 mg ibuprofen (diluted with 250 ml saline) will be administered 30 minutes before the end of surgery. All administrations will be applied through IV infusion over 30 minutes. Patients will be received tramadol with intravenous patient controlled analgesia (IV PCA) device during postoperative 24 hours. The PCA solution will be prepared with 500 mg tramadol in 100 mL of saline (5 mg/ml). The PCA device was adjusted as infusion: 2 ml/h, bolus: 2 ml, lockout period: 15 min.
  Other Names: Intravenous ibuprofen
  Arms: Intravenous ibuprofen

SUMMARY:
Primary aim of this prospective, randomized, double-blind clinical trial is to compare the analgesic effects of intravenous paracetamol and ibuprofen on postoperative pain, and secondary aim is the effects on tramadol consumption and side effects of tramadol in patients who underwent unilateral shoulder surgery.

DETAILED DESCRIPTION:
All surgical procedures are associated with acute pain and inflammation, with varying degrees of severity for patients, causing significant stress and discomfort. Effective postoperative pain management in shoulder surgery may reduce complications and improve postoperative care.

For postoperative pain, multimodal analgesic techniques are used to provide synergistic effects through different nociceptive mechanisms. Various analgesics are used for pain. Opioids, commonly used for postoperative pain, are the most popular drug group. Side effects such as sedation, respiratory depression, nausea-vomiting, pruritus and urinary retention that develop secondary to opioids may also be reduced by the combination of supplemental analgesics.

Adjuvant agents, including nonsteroidal anti-inflammatory drugs, may be used in combination with opioids. These drugs not only reduce pain but also control the underlying inflammatory process. In addition, combining nonsteroidal anti-inflammatory drugs and opioids can help to reduce the side effects by minimizing administration of total opioid consumption.

Intravenous paracetamol is an analgesic and antipyretic agent used as a first step drug for pain and fever control in adults and children. It has been clearly shown that intravenous paracetamol, with analgesic efficacy and good safety profile, reduces analgesic requirements for pain management. It provides better analgesic efficacy and reduces opioid consumption when used in combination with opioids.

Intravenous ibuprofen is the first and only intravenous nonsteroidal anti-inflammatory drugs approved in the United States for both pain and fever control in adults. It has been reported in multicenter studies that IV ibuprofen is safe and effective in postoperative pain management for orthopedic surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists scores 1-3
* 18-85 years

Exclusion Criteria:

* American Society of Anesthesiologists scores IV,
* Under the age of 18,
* Over the age of 85,
* Peptic ulcer disease,
* Hepatic and renal dysfunction,
* Severe cardiovascular and pulmonary disease,
* Allergic history to propofol, fentanyl, rocuronium, paracetamol, ibuprofen and tramadol,
* Emergency surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-04-09 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores | From end of anesthesia (15 minutes after anesthesia) to after 24 hours, up to 24 hours
  Visual Analog Scale (VAS, 0-10)

SECONDARY OUTCOMES:
Sedation score | From end of anesthesia (15 minutes after anesthesia) to after 24 hours, up to 24 hours
  Ramsey sedation score (1-6)
Tramadol consumption | From end of anesthesia (15 minutes after anesthesia) to after 24 hours, up to 24 hours
  Tramadol

CONTACTS AND LOCATIONS:
Overall Officials: Muhittin MD Calim, Study Director — Bezmialem Vakif University
Locations (1):
- Muhittin Calim, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tunali Y, Akcil EF, Dilmen OK, Tutuncu AC, Koksal GM, Akbas S, Vehid H, Yentur E. Efficacy of intravenous paracetamol and dexketoprofen on postoperative pain and morphine consumption after a lumbar disk surgery. J Neurosurg Anesthesiol. 2013 Apr;25(2):143-7. doi: 10.1097/ANA.0b013e31827464af. PMID 23360885